CLINICAL TRIAL: NCT00159471
Title: A Pilot Trial of Germline Polymorphisms as Predictors of Response to Gemcitabine, Docetaxel, and Capecitabine (GTX) in Metastatic or Unresectable Pancreatic Cancer.
Brief Title: Genes as Predictors of Response to Gemcitabine, Docetaxel, and Capecitabine (GTX) in Metastatic or Unresectable Pancreatic Cancer.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3P-03-2
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine, gemcitabine, docetaxel

SUMMARY:
This is a study for patients with advanced pancreatic cancer, using the drugs gemcitabine, docetaxel and capecitabine. Gemcitabine is a drug that has been approved by the FDA. Gemcitabine is been approved for treatment of cancer of the pancreas. It is also approved for treatment of lung cancer in combination with another drug called cisplatin. Docetaxel is a drug approved by the FDA. Docetaxel is approved for treatment of breast and lung cancer. Capecitabine is a drug approved by the FDA for treatment of cancer of the colon and rectum. This study will measure the levels of certain substances in participant's tumors. These substances (called genes, which are the cell's blueprint for these substances) affect how people's bodies react to the cancer drugs. Genes will also be measured in participant's blood. The purpose of this study is to see if these substances can predict survival and response in patients receiving the study drugs. In this study we wish to find out how long it takes for patients' cancers to worsen, and how long they survive after receiving the study drugs. The side effects of the combination of gemcitabine, docetaxel and capecitabine will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have clinically documented unresectable or metastatic pancreatic cancer and histologic confirmation of the diagnosis with tumor.
* Tissue from tumor must be available. This may be paraffin embedded tissue from previous biopsy/resection or if it is not available, a repeat biopsy must be performed.
* Patients must agree to have a 20 cc blood sample drawn in addition to routine labs with each cycle of chemotherapy.
* Patients must have measurable disease by clinical exam or radiologic studies, that is at least one lesion measurable in at least one dimension, measuring 20mm. If prior radiation therapy was administered, measurable disease must be outside the radiation field.
* Patients may have received prior adjuvant chemotherapy and/or radiation therapy; this must have been completed at least 6 months prior to the initiation of therapy for metastatic disease.
* Patients must have a Zubrod performance status of 0-2.
* Peripheral Neuropathy must be less than grade 1
* Patients must have a predicted life expectancy of at least 12 weeks.
* Patients must have a pre-treatment granulocyte count (i.e., segmented neutrophils + bands) of greater than 1,500/mm3, a hemoglobin level of greater than or equal to 9.0 gm/dl, and a platelet count of greater than 100,000/mm3.
* Patients must have adequate renal function as documented by a calculated creatinine clearance greater than 60.
* No major surgery within 1 month of starting study drug.

Exclusion Criteria:

* Patients who have received prior adjuvant therapy with more than one of the following agents: gemcitabine, docetaxel or capecitabine
* Patients who have received prior treatment for metastatic or unresectable pancreatic cancer.
* Patients may not have a history of an allergy to gemcitabine, taxanes or fluoropyrimidines and polysorbate 80.
* Patients with any active or uncontrolled infection, including known HIV infection.
* Patients with psychiatric disorders that would interfere with consent or follow-up.
* Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy.
* Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method while on treatment and for at least 3 months thereafter.
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis
* Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other anti-epileptic prophylaxis are ineligible.
* Patients with any other severe concurrent disease, which in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-02; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To see if patients with advanced pancreatic cancer treated with gemcitabine, docetaxel and capecitabine who bear more favorable genotypes of genes involved in drug metabolisms are more likely to have response and survive longer than those that do not.

SECONDARY OUTCOMES:
To assess time to progression, toxicity and to identify other molecular correlates of response, toxicity, and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C. / Norris Comprehensive Cancer Center
Locations (1):
- U.S.C / Norris Comprehensive Cancer Center, Los Angeles, California, United States